CLINICAL TRIAL: NCT00958386
Title: Open, Multicenter Phase II Study to Evaluate the Efficacy and Safety of the Combination of Panitumumab With Irinotecan in Patients With Wild-Type KRAS Metastatic Colorectal Cancer Refractory to Irinotecan Based Chemotherapy
Brief Title: Safety and Efficacy Study of Panitumumab+Irinotecan in Patients Wild-Type (WT) KRAS Metastatic Colorectal Cancer Refractory to Irinotecan Based Chemotherapy (SPECTRA)
Acronym: SPECTRA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spanish Cooperative Group for the Treatment of Digestive Tumours (TTD) (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TTD-08-06
Record Dates: First submitted 2009-08-12; First posted 2009-08-13 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Metastatic Colorectal Cancer
Keywords: colorectal cancer; Panitumumab; irinotecan
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Panitumumab+irinotecan
  Interventions: Drug: Panitumumab+irinotecan

INTERVENTIONS:
Drug: Panitumumab+irinotecan — Panitumumab will be administered as a 60 minute ± 15 minutes IV infusion, just prior to administration of chemotherapy at a dose of 6 mg/kg on day 1 of each cycle. A cycle of Panitumumab is defined as 14 days.
  Irinotecan chemotherapy (180 mg/m2 in 90 min on day 1 of each cycle) will be administered after the administration of Panitumumab.
  Each treatment cycle will have a duration of 14 days.

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of the combination of Panitumumab with Irinotecan in patients with Wild-Type KRAS metastatic colorectal cancer refractory to irinotecan based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Competent to comprehend, sign, and date an IEC-approved informed consent form.
* Men or women 18 years of age or older at the time the written informed consent is obtained.
* Histologically confirmed metastatic adenocarcinoma of the colon or rectum
* Wild-Type KRAS (No mutation) by allelic discrimination on tumor DNA.
* Karnofsky performance status ≥ 70% at the time of enrolment in the study.
* Within seven days prior to initiating study treatment:

  * Adequate bone marrow function: neutrophils ≥ 1.5x109/ L; platelets ≥ 100x109/L; hemoglobin ≥ 9g/dL.
  * Hepatic functions as follows: total bilirubin count ≤ 1.5 x ULN; ALAT and ASAT ≤ 2.5 x ULN (≤5 x ULN in case of liver metastasis).
  * Renal function: serum creatinine ≤1.5 ULN
  * Metabolic functions: magnesium ≥ lower limit of normal (LLN), calcium ≥ lower limit of normal (LLN)
* Life expectancy ≥ 3 months.

Exclusion Criteria:

* Prior malignant tumor in the last 5 years, except a history of basal cell carcinoma of the skin or pre-invasive cervical cancer.
* Unresolved toxicities from prior systemic therapy that, in the opinion of the investigator, does not qualify the patient for inclusion.
* Documented or suspected central nervous system metastases.
* Hormonal therapy, immunotherapy or experimental or approved proteins/antibodies (eg, Bevacizumab) ≤ 30 days before inclusion.
* Significant cardiovascular disease including unstable angina or myocardial infarction within 12 months before initiating study treatment or a history of ventricular arrhythmia.
* Prior anti-EGFr antibody therapy (eg, Cetuximab) or treatment small molecule EGFr tyrosine kinase inhibitors (eg, Erlotinib) or EGFR signal transduction inhibitors. Subjects who discontinue their first dose of anti-EGFR therapy (Cetuximab) because of an infusion reaction may participate in this clinical trial.
* Paraffin-embedded tissue or unstained tumor slides from primary or metastatic tumor not available (blocks available for Translational research).
* History of interstitial pneumonitis or pulmonary fibrosis or evidence of interstitial pneumonitis or pulmonary fibrosis on baseline chest CT scan.
* Treatment for systemic infection within 14 days before initiating study treatment.
* Acute or sub-acute intestinal occlusion and /or active inflammatory bowel disease or other bowel disease causing chronic diarrhoea (defined as > 4 loose stools per day).
* History of Gilbert's syndrome or dihydropyrimidine deficiency.
* History of any medical condition that may increase the risks associated with study participation or may interfere with the interpretation of the study results.
* Known positive test for human immunodeficiency virus infection, hepatitis C virus, and chronic active hepatitis B infection.
* Subject allergic to the ingredients of the study medication or to Staphylococcus protein A.
* Any co-morbid disease that would increase risk of toxicity.
* Any kind of disorder that compromises the ability of the subject to give written informed consent and/or comply with the study procedures.
* Any investigational agent within 30 days before initiation of the treatment.
* Subject who is pregnant or breast feeding.
* Surgery (excluding diagnostic biopsy or central venous catheter placement) and/or radiotherapy within 28 days prior to initiation of study treatment.
* Woman or man of childbearing potential not consenting to use adequate contraceptive precautions i.e. double barrier contraceptive methods (e.g. diaphragm plus condom), or abstinence during the course of the study and for 6 months after the last study drug administration for women, and 1 month for men.
* Subject unwilling or unable to comply with study requirements.
* Psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2009-08; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Objective response rate | 2009-2012

SECONDARY OUTCOMES:
disease control rate | 2009-2012
duration of response | 2009-2012
time to progression | 2009-2012
time to response | 2009-2012
time to treatment failure | 2009-2012
duration of stable disease | 2009-2012
Progression free survival | 2009-2012
Overall survival | 2009-2012
Safety profile | 2009-2012
Evaluation of molecular predictive markers | 2009-2012

CONTACTS AND LOCATIONS:
Overall Officials: Josep Tabernero, MD, phD, Study Chair — Hospital Vall de Hebrón. Barcelona. Spain; Enrique Aranda, MD; phD, Study Chair — Hospital Reina Sofía. Cordoba. Madrid
Locations (1):
- Spanish Cooperative Group for Gastrointestinal Tumour Therapy, Madrid, Spain